CLINICAL TRIAL: NCT01625494
Title: A Prospective Open-label Multicentre Study of Efficacy and Safety of Irbesartan/Amlodipine 4 Fixed Combination Therapy in Hypertensive Patients Uncontrolled on Irbesartan 150 mg or Amlodipine 5 mg Monotherapy
Brief Title: Study of Efficacy and Safety of Irbesartan/Amlodipine 4 Fixed Combination Therapy in Hypertensive Patients Uncontrolled on Irbesartan or Amlodipine Monotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRBES_L_05887; U1111-1117-9116 (Other: UTN)
Record Dates: First submitted 2012-06-19; First posted 2012-06-21 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2013-01

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Irbesartan; Amlodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Irbesartan/Amlodipine 150/5 mg fixed combination (Experimental): 1 tablet once daily in the morning for 4 weeks Patient will be first treated with irbesartan 150mg or amlodipine 5mg, 1 tablet /day for 4 weeks.
  If OBPM is controlled on monotherapy at week 4 (SBP <140 mmHg and DBP<90 mmHg), patient will be withdrawn from the study
  Interventions: Drug: Irbesartan/Amlodipine (150/5mg)
- Irbesartan/Amlodipine 150/10 mg fixed combination (Experimental): 1 tablet once daily in the morning for 4 weeks
  Interventions: Drug: Irbesartan/Amlodipine (150/10mg)
- Irbesartan/Amlodipine 300/5 mg fixed combination (Experimental): 1 tablet once daily in the morning for 4 weeks
  Interventions: Drug: Irbesartan/Amlodipine (300/5mg)
- Irbesartan/Amlodipine 300/10 mg fixed combination (Experimental): 1 tablet once daily in the morning for 4 weeks. If OBPM is controlled at week 12, patients will continue on the same therapy until the end of the study
  Interventions: Drug: Irbesartan/Amlodipine (300/10mg)

INTERVENTIONS:
Drug: Irbesartan/Amlodipine (150/5mg) — Pharmaceutical form: tablet Route of administration: oral
  Arms: Irbesartan/Amlodipine 150/5 mg fixed combination
Drug: Irbesartan/Amlodipine (150/10mg) — Pharmaceutical form: tablet Route of administration: oral
  Arms: Irbesartan/Amlodipine 150/10 mg fixed combination
Drug: Irbesartan/Amlodipine (300/5mg) — Pharmaceutical form: tablet Route of administration: oral
  Arms: Irbesartan/Amlodipine 300/5 mg fixed combination
Drug: Irbesartan/Amlodipine (300/10mg) — Pharmaceutical form:tablet Route of administration: oral
  Arms: Irbesartan/Amlodipine 300/10 mg fixed combination

SUMMARY:
Primary Objective:

- To assess the proportion of patients with controlled Office Blood Pressure Measurements (OBPM), defined as Systolic blood pressure < 140 mmHg and Diastolic blood pressure <90mmHg, at the end of the study

Secondary Objectives:

* To examine over time the antihypertensive effect of the 4 doses of the fixed combination therapy irbesartan/amlodipine on OBPM (SBP (systolic blood pressure) and DBP (diastolic blood pressure)
* To examine the proportion of patients with controlled OBPM (systolic BP<140 mm Hg and diastolic BP<90 mmHg) of the different dose groups over time
* To determine the incidence and severity of adverse events.

DETAILED DESCRIPTION:
16 weeks

* V1 (week 0): Inclusion visit.
* V2 (Week 4): Irbesartan/amlodipine 150/5 mg fixed combination visit
* V3 (Week 8): 1st dose escalation for patients in whom OBPM is not controlled (SBP ≥ 140 mmHg or DBP ≥ 90mmHg,
* V4 (Week 12): 2nd Dose escalation visit for patients in whom OBPM is not controlled (SBP ≥ 140 mmHg or DBP ≥ 90mmHg
* V5 (Week 16): End of study visit

ELIGIBILITY:
Inclusion criteria :

* Men and women ≥18 years old
* Established essential hypertension
* Treated with irbesartan 150 mg or amlodipine 5 mg as monotherapy for at least 2 weeks
* With uncontrolled systolic BP (blood pressure) defined as ≥140 mm Hg assessed by OBPM (office blood pressure measurements)
* Signed written informed consent obtained prior to inclusion to the study

Exclusion criteria:

* Mean systolic BP ≥180 mm Hg and/or mean diastolic BP ≥110 mm Hg by OBPM on Visit 1
* Known or suspected causes of secondary hypertension
* Patients with bilateral artery stenosis, renal artery stenosis in a solitary kidney, renal transplant or only has one functioning kidney
* Known contraindications or hypersensitivity to either amlodipine or irbesartan or to the combination
* History of angioedema related to the administration of an angiotensin II receptor antagonist or any combination of the drugs used
* Severe hepatic impairment (Alanine aminotransferase (ALT) or Aspartate aminotransferase (AST) >5 times the upper normal limit (ULN) or history of hepatic encephalopathy, esophageal varices or portocaval shunt)
* Severe renal impairment (glomerular filtration rate <30 ml/min)
* Concomitant use of any other antihypertensive treatment except of Irbesartan and Amlodipine
* Administration of any other investigational drug within 30 days before inclusion
* Presence of any other conditions that would restrict or limit the patient participation for the duration of the study
* Pregnant or breast feeding women
* Women of childbearing potential unable or unwilling to use an acceptable method to avoid pregnancy for the entire study period
* Patient is the investigator or any sub-investigator, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the protocol

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2012-05; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with controlled OBPM (SBP<140 mmHg and DBP<90 mmHg) at the end of the study | up to 16 weeks

SECONDARY OUTCOMES:
Proportion of patients with controlled OBPM by visit and treatment group | up to 16 weeks
  at Visit 3 (Week 8), at Visit 4 (Week 12) and at Visit 5 (Week 16)
Mean change in OBPM between 2 visits | up to 16 weeks
  Visit 2 (Week 4) and Visit 5 (Week 16), Visit 2 (Week 4) and Visit 4 (week 12), Visit 2 (Week 4) and Visit 5 (Week 16), Visit 3 (Week 8) and Visit 4 (Week 12), Visit 3 (Week 8) and Visit 5 (Week 16)
Number of patients with adverse events | up to 16 weeks
Number of patients who discontinue from the study due to adverse events | up to 16 weeks
Number of patients with abnormal liver function | up to 16 weeks
  As measured by AST, ALT, total bilirubin and serum creatinine

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Moscow, Russia